CLINICAL TRIAL: NCT03125226
Title: TraceIT TM Hydrogel Tissue Marker for Patients Receiving Definitive Chemoradiation for Bladder Cancer
Brief Title: TracelT Hydrogel in Localizing Bladder Tumors in Patients Undergoing Radiation Therapy for Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Zeng, Associate Professor, Department of Radiation Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9798; NCI-2017-00525 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9798 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG3117001 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (TracelT hydrogel) (Experimental): Patients undergo transurethral resection of bladder tumors and receive TracelT hydrogel via injection. Patients undergo standard of care radiation therapy within 8 weeks of TracelT hydrogel placement.
  Interventions: Device: Polyethylene Glycol Hydrogel

INTERVENTIONS:
Device: Polyethylene Glycol Hydrogel — Given TracelT hydrogel via injection
  Other Names: PEG Hydrogel

SUMMARY:
This pilot clinical trial studies how well TracelT hydrogel works in localizing bladder tumors in patients undergoing radiation therapy for bladder cancer. TracelT hydrogel marks the location of a bladder tumor and makes it more visible during imaging tests. Using TracelT hydrogel tissue marker may help doctors learn more about tumor location and altering radiation dosage for bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To utilize the TraceIT hydrogel tissue marker in localizing bladder tumors during transurethral resection of bladder tumors (TURBT).

II. To improve identification of gross tumor or tumor bed location in patients receiving chemoradiation treatment for bladder cancers.

SECONDARY OBJECTIVES:

I. To report adverse events surrounding the placement of the TraceIT tissue marker.

II. To calculate the actual dose received by the bladder tumor bed, as delineated by the hydrogel.

III. To compare the dosimetric impact to the tumor bed of daily patient alignment to the pelvic bones, versus alignment to the whole bladder, versus alignment to the hydrogel markers.

IV. To calculate the amount of normal tissue radiation dose decrease achievable without losing tumor coverage, with better tumor targeting with hydrogel placement.

OUTLINE:

Patients undergo transurethral resection of bladder tumors and receive TracelT hydrogel via injection. Patients undergo standard of care radiation therapy within 8 weeks of TracelT hydrogel placement.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy of the bladder
* No prior cystectomy
* Treatment plan for bladder must include at least 4 weeks of daily radiation treatment (most patients will receive chemotherapy concurrent with radiation, but this is not required for trial enrollment)
* Patient must undergo TraceIT hydrogel placement within 8 weeks prior to starting radiation therapy for bladder cancer
* Participants must have a complete history and physical examination within 60 days of study entry
* Participants must be able to provide informed consent for treatment and trial participation
* No restrictions on prior treatment to be eligible

Exclusion Criteria:

* Prior cystectomy
* Unable to have TraceIT hydrogel placement < 8 weeks prior to beginning radiation treatment
* Treatment for metastatic bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (TracelT Hydrogel)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 73 [53 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Interfraction Motion of the Marker Measured by Cone Beam Computed Tomography (CT) and x/y/z Coordinates
Description: Daily changes will be compared across the patient group as well as within each subjects' treatment course.
Time Frame: Baseline up to 8 weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
cm | 0.62 (0.54)
Statistical Analysis 1: Comparison: Supportive Care (TracelT Hydrogel); Coordinates in x/y/z planes were assigned to each hydrogel marker on the planning CT and daily CBCT to calculate interfraction motion; Test type: Other — Single group mean and standard deviation; Single group mean and standard deviation

2. Primary Outcome: Changes in Tumor Bed Size and Shape as Delineated by the Hydrogel and Measured by Cone Beam CT and x/y/z Coordinates
Description: Daily changes will be compared across the patient group as well as within each subjects' treatment course. These changes will be tracked during the entire radiation course (typically 4-8 weeks), yielded a distribution of x/y/z positions for each patient.
Time Frame: Baseline up to 8 weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
cm | 0.21 (0.48)

3. Secondary Outcome: Daily Dose of Radiation to the PTV as Based on Alignment to the Hydrogel Location Versus Alignment to Whole Bladder Location Versus Alignment to Bony Antonym
Description: Daily pre-radiation imaging will be used to run the radiation treatment plan, to calculate the daily dose to the PTV based on alignment to the hydrogel location, versus alignment to whole bladder location, versus alignment to bony anatomy.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Error); unit: percentage of total dose
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
percentage of total dose | 95 (2)

4. Secondary Outcome: Daily Dose to the Planning Tumor Volume (PTV) Based on Hydrogel Location
Description: Daily pre-radiation imaging will be used to run the radiation treatment plan, to calculate the daily dose to the PTV based on hydrogel location. Total radiation dose to the PTV can then be calculated as the sum of the daily dose.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Error); unit: percentage of total dose
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
percentage of total dose | 99 (2)

5. Secondary Outcome: Number of Participants With Adverse Events Caused by Hydrogel
Description: Graded by the Common Terminology Criteria in Adverse Events version 4.0
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
Participants | 0

6. Secondary Outcome: Smallest Setup Margin Required for Consistent Coverage of the Gross Tumor Volume (GTV)
Description: Daily pre-radiation imaging will be used to identify the smallest setup margin required for consistent coverage of the GTV, which is likely smaller than the current standard of care setup margin of at least 2 cm around the GTV.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Supportive Care (TracelT Hydrogel)
Number analyzed (Participants) | 12
mm | 10 (3)
Statistical Analysis 1: Comparison: Supportive Care (TracelT Hydrogel); Test type: Other — The Van Herk (VH) margin equation for the planning target volume margin, as a function of systemic and random errors, was calculated such that the CTV receives at least 95%-prescription dose in 90% of patients; The Van Herk (VH) margin equation for the planning target volume margin, as a function of systemic and random errors, was calculated such that the CTV receives at least 95%-prescription dose in 90% of patients

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Supportive Care (TracelT Hydrogel)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (TracelT Hydrogel) (N=12)
Urinary frequency (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03125226/Prot_SAP_000.pdf